CLINICAL TRIAL: NCT05948995
Title: Comparison Between Abduction External Rotation Brace and Arm Sling After Arthroscopic Rotator Cuff : A Randomized Controlled Trial
Brief Title: Comparison Between Abduction External Rotation Brace and Arm Sling After Arthroscopic Rotator Cuff
Acronym: ARCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 022/2566
Record Dates: First submitted 2023-06-29; First posted 2023-07-17 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Arthroscopic Rotator Cuff Repair

STUDY DESIGN:
Intervention Model Description: The participants were randomly divided into two groups. The control group received arm sling post operative arthroscopic rotator cuff repair. The experimental group received abduction external rotation brace post operative arthroscopic rotator cuff repair.
Who Masked: Outcomes Assessor
Masking Description: On the follow up date , both groups will be removed sling / brace before receiving by outcome assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm sling (No Intervention): Conventional arm sling Arm position : Internal rotation , Adduction
- Abduction external rotational brace (Experimental): Abduction external rotational brace Arm position : Abduction , External rotation
  Interventions: Device: Abduction external rotation brace

INTERVENTIONS:
Device: Abduction external rotation brace — Abduction external rotation brace Arm position : Abduction , External rotation
  Other Names: Arm sling with abduction pillow
  Arms: Abduction external rotational brace

SUMMARY:
Comparison between Abduction External Rotation Brace and Arm Sling after Arthroscopic Rotator Cuff : A Randomized Controlled Trial Comparison of primary outcome : range of motion (at pre-operative , post-operative) , pain score , shoulder functional score

DETAILED DESCRIPTION:
Comparison between Abduction External Rotation Brace and Arm Sling after Arthroscopic Rotator Cuff : A Randomized Controlled Trial Comparison of primary outcome : range of motion (at pre-operative , post-operative) , pain score , shoulder functional score There are gaps of knowledge which sling/brace are the best for post operative arthroscopic rotator cuff repair Because patient who underwent arthroscopic rotator cuff repair have to wear these sling/brace for at least 1 month after operation , the better one could reduce post-operative shoulder stiffness , decrease pain and improve functional shoulder score

ELIGIBILITY:
Inclusion Criteria:

* Patient with full thickness rotator cuff tear
* Plan for arthroscopic rotator cuff repair

Exclusion Criteria:

* Revision cuff surgery
* Unable to answer question
* Previous shoulder surgery
* Full thickness subscapularis tear

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of range of motion of shoulders from baseline | At postoperative 3 weeks
  Measurement by Goniometer into degrees (forward flexion, external rotation, internal rotation)
Change of range of motion of shoulders from baseline | At postoperative 6 weeks
  Measurement by Goniometer into degrees (forward flexion, external rotation, internal rotation)
Change of range of motion of shoulders from baseline | At postoperative 3 months
  Measurement by Goniometer into degrees (forward flexion, external rotation, internal rotation)
Change of range of motion of shoulders from baseline | At postoperative 6 months
  Measurement by Goniometer into degrees (forward flexion, external rotation, internal rotation)
Change of range of motion of shoulder from baseline | At postoperative 1 year
  Measurement by Goniometer into degrees (forward flexion, external rotation, internal rotation)

SECONDARY OUTCOMES:
Change of visual analog scale for pain from baseline | Change from visual analog scale after 6 weeks postoperative
  Range from 1-10 (1 = minimum pain, 10 = maximum pain)
Change of constant Murley's score from baseline | Change from visual analog scale after 6 weeks postoperative
  Score 0-100 (Functional shoulder score), 0 = worst, 100 = best
Change of the Thai version of the Shoulder Pain and Disability Index from baseline | Change from visual analog scale after 6 weeks postoperative
  Thai functional shoulder score 0 = worst, 100 = best

CONTACTS AND LOCATIONS:
Overall Officials: Chuenrutai Yeekian, Ph.D., Study Chair — QSMVH
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Si Racha, Thailand

IPD SHARING:
Plan to Share IPD: No
Data was save in form of microsoft excel spreadsheet and SPSS file